CLINICAL TRIAL: NCT06806150
Title: The INSPIRE Study: INvestigation of Swiss Physicians Inner-life, Resilience, and Emotions
Acronym: INSPIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2023-00963
Record Dates: First submitted 2025-01-31; First posted 2025-02-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Burnout, Professional; Emotional Exhaustion; Emotions; Wellness, Psychological; Satisfaction, Personal
Keywords: Psychological resilience; Positive Psychology
MeSH Terms: conditions — Burnout, Professional; Emotional Exhaustion; Psychological Well-Being; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants: Control participants are aware of the trial but do not know they are assigned to the control arm, as they are treated as part of the larger cohort and do not receive the intervention.
  Investigators: Investigators are masked because recruitment and assignment are automated, ensuring they do not know which participants are in the intervention or control arms.
  Outcome Assessors: Researchers analyzing the data remain blinded to group allocation to minimize bias in data interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 - General Positive Psychology Reflection (Experimental): Participants engage in an 8-day web-based intervention involving positive psychology exercises focused on general life situations.
  Interventions: Behavioral: INSPIRE Life Reflection
- Intervention 2 - Work-Specific Positive Psychology Reflection (Experimental): Participants engage in the same 8-day web-based intervention, but the focus is specifically on positive reflections related to work and patient interactions.
  Interventions: Behavioral: INSPIRE Work Reflection
- Control group (No Intervention): Participants complete assessments but do not receive the intervention.

INTERVENTIONS:
Behavioral: INSPIRE Life Reflection — An 8-day web-based positive psychology intervention encouraging participants to reflect on positive aspects of their daily lives. Activities include gratitude exercises, self-compassion writing, and recognizing meaningful moments.
  Arms: Intervention 1 - General Positive Psychology Reflection
Behavioral: INSPIRE Work Reflection — An 8-day web-based positive psychology intervention encouraging participants to reflect on positive aspects of their work experiences. Activities include gratitude exercises, self-compassion writing, and recognizing meaningful professional interactions.
  Arms: Intervention 2 - Work-Specific Positive Psychology Reflection

SUMMARY:
The goal of this clinical trial, nested within an observational cohort study, is to evaluate whether two positive psychology web-based interventions can reduce emotional exhaustion and improve overall well-being in practicing physicians in Switzerland. The main questions it aims to answer are:

Does participation in positive psychology interventions reduce emotional exhaustion at three months post-intervention? How do these interventions impact physician wellness, job satisfaction, comfort with end-of-life communication and other aspects of physicians' emotional well-being?

Researchers will compare the effects of two intervention arms (general reflection vs. work-specific reflection) to a control group to determine whether focusing on work-specific aspects leads to greater improvements in emotional exhaustion and job-related outcomes.

Participants will:

* Complete an 8-day intervention consisting of positive psychology activities delivered online.
* Complete baseline and follow-up assessments over the study period

DETAILED DESCRIPTION:
Burnout, emotional exhaustion, and moral distress are widespread among physicians, negatively impacting patient care, job satisfaction, and physician retention in the workforce. While interventions targeting burnout exist, many require significant time commitments or institutional support, limiting accessibility.

Positive psychology interventions, which emphasize strengths-based approaches such as self-reflection, gratitude, and self-compassion, have shown promise in enhancing resilience and well-being.

The INSPIRE study is a randomized controlled trial (RCT) nested within an observational cohort using a Trial within Cohort (TwiC) design. It evaluates two web-based positive psychology interventions aimed at reducing emotional exhaustion and improving physician well-being.

A subset of cohort participants is randomized into one of three arms: a control group, a general life reflection intervention, or a work-focused reflection intervention. The interventions consist of an 8-day structured self-reflection program delivered online.

The study employs automated randomization, triple masking (participants, investigators, and outcome assessors), and longitudinal assessments over one year. Findings will inform the scalability of low-burden interventions for physician burnout prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Be a practicing physician in Switzerland
2. Working at least 40% in a clinical capacity
3. Be willing and able to provide informed consent
4. Expecting to be professionally active until 2028

Exclusion Criteria:

1. Retired physician or physician seeking retirement within 3 years from first participation in the study
2. Physician unable to participate in one of the study languages: English, German, or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to all gender identities, including male, female, non-binary, and those who prefer not to disclose it.
Enrollment: 450 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Emotional Exhaustion | 3 months post-intervention
  Emotional Exhaustion subscale of the MBI-HSS

SECONDARY OUTCOMES:
Change in Emotional Exhaustion | Baseline to 2 weeks, 1 month, 6 months, 1 year
  Emotional Exhaustion subscale of the MBI-HSS
Change in Depersonalization | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  Depersonalization subscale of the MBI-HSS
Change in Personal Accomplishment | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  Personal accomplishment subscale of the MBI-HSS
Change in Physician wellbeing | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  Physician Wellness Inventory (PWI)
Change in Job Satisfaction | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  Physician Job Satisfaction Scale
Change in comfort with End-of-Life Communication | Baseline to 1 month, 3 months, 6 months, 1 year
  Communication about End of Life Survey
Change in Mindfulness | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  Mindful Attention Awareness Scale (MAAS-Trait)
Change in Compassionate Care | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  Santa Clara Brief Compassion Scale
Change in Emotion Regulation | Baseline to 1 month, 3 months, 6 months, 1 year
  Emotion Regulation Questionnaire (ERQ)
Change in Positive and Negative Affect | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  Positive and Negative Affect Schedule (PANAS)
Change in Authenticity | Baseline to 3 months, 6 months, 1 year
  Inauthenticity Scale
Resilience | Baseline to 2 weeks, 1 month, 3 months, 6 months, 1 year
  2-item Connor-Davidson resilience scale

OTHER OUTCOMES:
Perceived impact of the INSPIRE Interventions | Within 6 months post-intervention
  Qualitative interviews with a subset of trial participants to understand perceived impact of the INSPIRE interventions.
Acceptability of the INSPIRE Interventions | Within 6 months post-intervention
  Qualitative interviews with a subset of trial participants to understand acceptability of the INSPIRE interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia C Zambrano, PhD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available for research purposes upon request. Data will include survey responses and outcome measures but will exclude any personally identifiable information
Time Frame: 18 months after publication of primary results and will remain accessible for at least 5 years
Access Criteria: Researchers can request access by submitting a proposal to the study investigators. Access will be granted to qualified researchers for scientifically valid analyses, subject to data-sharing agreements and ethical considerations.